CLINICAL TRIAL: NCT02545777
Title: The Clinical Study on Treating Acute Gouty Arthritis Using Both Internal and External Therapy of Tonifying Spleen and Descending Turbid
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Wang Shidong, Beijing University of Chinese Medicine, Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-ZYLC-001
Record Dates: First submitted 2015-09-02; First posted 2015-09-10 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Acute Gouty Arthritis
Keywords: Acute gouty arthritis; tonifying spleen and descending the turbid; soaking; wet wrapping

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- treatment group (Active Comparator): Take oral medicine of tonifying spleen and descending turbid, one bag each time, two times a day, continuous treatment for 10 days.The onset of the joints afford steeping washing and wet wrapping medicine of descending turbid and clearing heat, once per day, continuous treatment for 10 days.
  Interventions: Drug: Oral medicine of tonifying spleen and descending turbid; Drug: Steeping and washing medicine of descending turbid and clearing heat; Drug: Wet wrapping medicine of descending turbid and clearing heat
- Control group (Active Comparator): Take diclofenac sodium enteric-coated, 50 mg, three times a day, continuous treatment for 10 days.
  Interventions: Drug: diclofenac sodium enteric-coated

INTERVENTIONS:
Drug: diclofenac sodium enteric-coated
  Arms: Control group
Drug: Oral medicine of tonifying spleen and descending turbid — Ingredient:cortex phellodendrine, rhizoma atractylodis, radix cyathula, coix seed, cotton Bi Xie,rhizoma smilacis glabrae
  Arms: treatment group
Drug: Steeping and washing medicine of descending turbid and clearing heat — Ingredient: turmeric, rhubarb, cortex phellodendrine, rhizoma atractylodis, rhizoma arisaema, angelica dahurica,garden balsam stem, pseudobulbus cremastrae seu pleiones
  Arms: treatment group
Drug: Wet wrapping medicine of descending turbid and clearing heat — Ingredient:turmeric, rhubarb, cortex phellodendrine, rhizoma atractylodis, rhizoma arisaema, angelica dahurica, pseudobulbus cremastrae seu pleiones.
  Arms: treatment group

SUMMARY:
This research is based on spleen trapped by dampness and turbid which is the pathogenesis of gouty arthritis.It uses effective prescription of Endocrinology of Dongzhimen Hospital.In this study, the investigators use multi-center randomized parallel controlled clinical trials.The treatment groups are afforded oral traditional Chinese medicine decoction-tonifying spleen and descending the turbid decoction as well as soaking and wet wrapping.The control groups are afforded diclofenac sodium enteric-coated tablets as a positive control drug.The outcome is evaluated by condition of symptoms remission,pain relief time, recurrence rate and laboratory index to determine the efficacy of internal and external treatment.And the research will provide optimized diagnosis and treatment program. The investigators hope this research will also get tonifying spleen and descending the turbid internal and external treatment for gouty arthritis effective clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75, and gender unlimited;
2. The patients must meet western medicine diagnostic criteria for acute gouty arthritis;
3. The patients must meet that integral syndrome differentiation conforms to the spleen beset by dampness syndrome and local syndrome differentiation conforms to blockage disease due to heat.

Exclusion Criteria:

1. Secondary hyperuricemia, such as cancer and perichemotherapy of leukemia, renal failure, cirrhosis of the liver and drug effect(such as diuretics, aspirin, antitubercular agents), et al.
2. Acute infectious diseases, stroke, acute myocardial infarction ,as well as other acute diseases and tumors, rheumatoid arthritis.
3. Patients with peptic ulcer and gastrointestinal bleeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The relief of symptoms | After take the drug 10 days
  This measure is a composite outcome according to the joint red and swollen, joint pain, and restricted movement(Excellent:Complete resolution of symptoms, joint function returning to normal. The score of joint pain, joint red and swollen and joint motion is 0.Effective:The main symptoms mostly disappear. Joint function is improvement, but still have the joint red,swollen,pain and limited activity.Invalid: There is no improvement compared with before treatment).The unit of measure is scale.
The gout relief index | After take the drug 10 days
  The gout relief index = [gout relief time (days) ÷ 10 (days)] x 100%.The unit of measure is scale.
Compare scores of syndrome before treatment and after it. | After take the drug 10 days
  Using nimodipine method: nimodipine = [(scores of syndrome before treatment minus score after it) ÷scores of syndrome before treatment] x 100%.The unit of measure is scale.

SECONDARY OUTCOMES:
Recurrence rate | Following up for 1 month
  Recurrence rate=number of patient recurring acute gouty arthritis ÷total cases of each group.The unit of measure is number.
Recurrence time | Following up for 1 month
  Compare the days of cases recurring acute gouty arthritis of each group.The unit of measure is days.
The dosage of colchicine of two groups in observation period | After take the drug 10 days
  The unit of measure is mg.
Blood uric acid before and after the treatment. | After take the drug 10 days
White blood cell count before and after the treatment. | After take the drug 10 days
Erythrocyte sedimentation rate before and after the treatment. | After take the drug 10 days

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - No.3 Hospital Affiliated to Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Dongzhimen Hospital Affiliated to Beijing University of Chinese Medicine, Beijing, Beijing Municipality